CLINICAL TRIAL: NCT01365754
Title: Posterior Dynamic Stabilization Versus Fusion in the Treatment of Lumbar Degenerative Disease
Brief Title: Dynamic Stabilization Versus Fusion
Acronym: DYNORFUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYN-1009-MEY-0000-I
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
Keywords: Lumbar degenerative disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): A - Fusion
  Interventions: Procedure: standard
- B (Active Comparator): B - Dynamic (new)
  Interventions: Procedure: new

INTERVENTIONS:
Procedure: standard — fusion
  Arms: A
Procedure: new — dynamic stabilization
  Arms: B

SUMMARY:
The purpose of this study is to compare posterior dynamic stabilization with fusion in the treatment of lumbar degenerative disease.

DETAILED DESCRIPTION:
Two strategies for treatment of degenerative lumbar instability are in frequent clinical use: fusion versus dynamic stabilization. Up to now it is not clear whether fusion (Gold-standard) or the non-fusion technique is superior. Nevertheless some data are available that dynamic stabilization as a less invasive technique can achieve similar or better results concerning patient satisfaction and re-OP rate compared with fusion as the standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Mono- or bisegmental symptomatic lumbar degenerative disease with or without stenosis
* Indication for fusion with (i) spondylolisthesis of at least 5mm or segmental vertebral motion of at least 3mm or 10º on flexion/extension radiographs, (ii) predominant low back pain in combination with Modic changes
* Failure of adequate conservative measures for more than 3 months
* Correctly signed informed consent form

Exclusion Criteria:

* Olisthesis more than grade I, spondylolisthesis vera, spondylolysis without olisthesis or spinal deformity (i.e. scoliosis of more than 20°, sagittal imbalance)
* Significant comorbidity impeding with surgical success (e.g. osteoporosis, rheumatoid arthritis, mental illness)
* Previous fusion or stabilization surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Difference in Oswestry disability index (ODI) between treatment groups at 2 years post intervention | 2 years after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. med. Bernhard Meyer, München, Germany